CLINICAL TRIAL: NCT07295366
Title: Early Administration of PCSK9 Inhibitors After Thrombectomy for Atherosclerotic Acute Ischemic Stroke: A Randomized Controlled Trial
Acronym: EPOCH-TECT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XYFY2025-KL574-01
Record Dates: First submitted 2025-12-07; First posted 2025-12-19 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Acute Stroke
Keywords: Acute Ischemic Stroke; Mechanical Thrombectomy; Atherosclerosis; PCSK9 Inhibitor; Early Neurological Deterioration
MeSH Terms: conditions — Stroke; Ischemic Stroke; Atherosclerosis | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Intervention Group: Thrombectomy alone + evolocumab
  Thrombectomy alone: Mechanical thrombectomy performed according to guidelines (may include necessary angioplasty/stent implantation).
  Elavolocumab: 420 mg subcutaneously injected within 6 hours after recanalization (140 mg x 3 injections, pre-filled 3 mL total), at the location of the abdomen, lateral thigh, or lateral upper arm.
  Both groups received standardized drug therapy: antithrombotic/lipid-regulating/blood pressure/blood glucose/fluid management and rehabilitation: in accordance with the latest clinical guidelines.
  Interventions: Drug: Elavolocumab(420 mg injections)
- control group (No Intervention): Control group: simple thrombectomy
  Both groups received standardized drug therapy: antithrombotic/lipid-regulating/blood pressure/blood glucose/fluid management and rehabilitation: in accordance with the latest clinical guidelines.

INTERVENTIONS:
Drug: Elavolocumab(420 mg injections) — Intervention Group: Thrombectomy alone + evolocumab Thrombectomy alone: Mechanical thrombectomy performed according to guidelines (may include necessary angioplasty/stent implantation). Elavolocumab: 420 mg subcutaneously injected within 6 hours after recanalization (140 mg x 3 injections, pre-filled 3 mL total), at the location of the abdomen, lateral thigh, or lateral upper arm.
  Arms: intervention group

SUMMARY:
This study (EPOCH-TECT) was a single-center, randomized, open-label, blinded, endpoint-assessing controlled trial conducted at the Affiliated Hospital of Xuzhou Medical University. It aimed to investigate the efficacy and safety of administering the PCSK9 inhibitor evolocumab early (within 6 hours) after successful thrombectomy in patients with atherosclerotic large vessel occlusive stroke. The study planned to enroll 60 patients, who were randomly assigned 1:1 to either the "thrombectomy + evolocumab" group or the "thrombectomy alone" group. The primary endpoint was the incidence of early neurological deterioration within 7 days post-procedure (NIHSS score increase ≥2 points from post-operative best or death from any cause); secondary endpoints included 24-hour recanalization failure rate, 90-day functional recovery (mRS score 0-2), changes in serum biomarkers, and safety indicators such as symptomatic intracranial hemorrhage. This study aimed to provide prospective evidence for early intensive lipid-lowering and neuroprotective strategies after thrombectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-85 years old, gender not limited, gender ratio not limited.
2. The clinical diagnosis was acute ischemic stroke with occlusion of the anterior circulation large vessels. CTA/DSA confirmed that the responsible vessel for this stroke occlusion was located in the intracranial segment of the internal carotid artery and the M1 segment of the middle cerebral artery.
3. The time from onset to puncture is within 24 hours, and the patient receives mechanical thrombectomy (MT) (including direct thrombectomy and intravenous thrombolysis bridging thrombectomy), with postoperative vascular recanalization reaching mTICI grade 2b or 3. The surgical indications and time window follow the current guidelines and imaging criteria of key randomized controlled trials (RCTs). The definitions are as follows: Early window (0-6 h): Meeting the usual EVT indications (anterior circulation LVO, baseline NIHSS ≥ 6, ASPECTS ≥ 6, or center-defined criteria), the interventional team decides to perform MT; Late window (6-24 h): Meeting one of the imaging selection criteria of DAWN or DEFUSE-3 (based on CTP-RAPID or MRI-DWI/perfusion):

   ·DAWN (6-24 h) (any one): Age ≥ 80 years: NIHSS ≥ 10 and core infarct volume < 21 mL; Age < 80 years: NIHSS ≥ 10 and core < 31 mL; Age < 80 years: NIHSS ≥ 20 and core 31-51 mL.

   • DEFUSE-3 (6-16 h) (all conditions must be met): Core <70 mL, mismatch ratio (penumbra/core) ≥1.8, mismatch volume ≥15 mL, and Tmax >6 s volume >15 mL.
4. The etiological classification is intracranial arteriosclerosis-LAA (ICAD-LAA). The definition is as follows: imaging evidence supports the presence of atherosclerotic stenosis/plaque in the responsible vessel (such as severe stenosis/occlusion of the proximal internal carotid artery or middle cerebral artery) and the patient has corresponding underlying atherosclerosis (such as other intracranial/extracranial artery stenosis, hypertension, diabetes, etc.).
5. Baseline National Institutes of Health Stroke Scale (NIHSS) score ≥ 6 points.
6. Before the onset of the disease, the patient had good daily living abilities and an mRS score ≤ 2 (no severe disability).
7. Able to complete the injection of research drugs as required.
8. The patient or his or her legal representative shall sign a written informed consent form, understand the research content and agree to cooperate with the follow-up.

Exclusion Criteria:

1. Non-atherosclerotic lesions (such as arterial dissection, Moyamoya disease, vasculitis, embolism of unknown origin, etc.).
2. Patients who present with significant intracranial hemorrhage or excessively large cerebral infarction volume upon admission, making them unsuitable for continued participation in the study.
3. The cause of stroke is cardioembolism (such as a history of heart disease such as atrial fibrillation or valvular heart disease).
4. Individuals with a clear history of allergy to evolocumab or its excipients.
5. Patients with severe liver and kidney dysfunction: baseline alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3 times the upper limit of normal, or significantly reduced creatinine clearance (eGFR < 30 mL/min/1.73m²).
6. Patients with active severe infection, immune system disease or other serious comorbidities that may significantly affect prognosis (such as active tumors, terminal diseases, etc.).
7. Patients who have been treated with PCSK9 inhibitors within the past 4 weeks (to avoid affecting the study due to changes in tolerance or mechanism of action).
8. Pregnant or lactating women.
9. Expected survival <90 days or accompanied by other serious diseases.
10. Currently participating in other interventional clinical studies.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-18 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Early deterioration of neurological function (END) | Within 7 days post-thrombectomy
  The incidence of early neurological deterioration (END) within 7 days, defined as an increase of ≥2 points in NIHSS score compared to the best post-procedure level or death from any cause.
Incidence of symptomatic intracranial hemorrhage (sICH) within 90 days, defined according to the Heidelberg Bleeding Classification criteria. | Within 90 days post-thrombectomy
  Incidence of symptomatic intracranial hemorrhage (sICH) within 90 days, defined according to the Heidelberg Bleeding Classification criteria.

OTHER OUTCOMES:
Ineffective reperfusion rate at 24-36 hours post-procedure | Within 24-36 hours post-procedure
  Ineffective reperfusion rate observed by CTA+CTP re-examination at 24-36 hours post-procedure
Change in NIHSS score between baseline (Day 0) and Day 7 | within 1-7 days post-procedure
  Change in NIHSS score from post-procedure Day 0 to Day 7
Proportion of patients with mRS 0-2 at 90 days | Within 90 days post-thrombectomy
  Proportion of patients with mRS 0-2 at 90 days
Incidence of new ischemic stroke at 90 days | Within 90 days post-thrombectomy
  Incidence of new ischemic stroke at 90 days
EQ-5D-5L health-related quality of life score at 90 days | Within 90 days post-thrombectomy
  EQ-5D-5L health-related quality of life score at 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Yu Feng, MD, PhD, Principal Investigator — The Affiliated Hospital of Xuzhou Medical University; Yanbo Cheng, MD, PhD, Study Director — The Affiliated Hospital of Xuzhou Medical University
Locations (1):
- Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
Participants do not consent to the data sharing about themselves. IPD involves privacy and ethical issues.